CLINICAL TRIAL: NCT03650114
Title: An Open-label, Single Arm, Multi-center Extension Study Evaluating Long-term Safety, Tolerability and Effectiveness of Ofatumumab in Subjects With Relapsing Multiple Sclerosis
Brief Title: Long-term Safety, Tolerability and Effectiveness Study of Ofatumumab in Patients With Relapsing MS
Acronym: ALITHIOS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMB157G2399; 2023-507906-15 (Other: EU CTIS)
Record Dates: First submitted 2018-08-17; First posted 2018-08-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: ofatumumab; relapsing multiple sclerosis
MeSH Terms: interventions — ofatumumab; Tetanus Toxoid; keyhole-limpet hemocyanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Subcutaneous injection
  Interventions: Biological: Ofatumumab; Biological: Tetanus toxoid (TT) containing vaccine (Td, Tdap); Biological: 13-valent pneumococcal conjugate vaccine (13-PCV); Biological: 23-valent pneumococcal polysaccharide vaccine (23-PPV); Biological: Seasonal Quadrivalent influenza vaccine; Biological: Keyhole limpet hemocyanin (KLH) neo-antigen

INTERVENTIONS:
Biological: Ofatumumab — subcutaneous injection of 20 mg ofatumumab every 4 weeks
Biological: Tetanus toxoid (TT) containing vaccine (Td, Tdap) — 0.5mL Vial/Syringe Containing 5 limit of flocculation (LF) tetanus toxoid
Biological: 13-valent pneumococcal conjugate vaccine (13-PCV) — 0.5mL Vial/Syringe
Biological: 23-valent pneumococcal polysaccharide vaccine (23-PPV) — 0.5mL Vial/Syringe
Biological: Seasonal Quadrivalent influenza vaccine — Seasonal 2020-2021 0.5mL Vial/Syringe (trivalent may be used where quadrivalent is not available)
Biological: Keyhole limpet hemocyanin (KLH) neo-antigen — 1mg Vial

SUMMARY:
The purpose of this study is to collect long-term safety, tolerability, effectiveness and health outcomes data in eligible subjects who have participated in a Novartis ofatumumab clinical MS study.

Vaccination sub-study The purpose of this research sub-study is to find out the effects of ofatumumab on the development of antibody responses to selected vaccines and keyhole limpet hemocyanin (KLH) neo-antigen in subjects with relapsing multiple sclerosis (RMS).

COVID-19 sub-study:

The purpose of this research sub-study is to explore the immune response following Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) vaccination in a subset of subjects on long-term ofatumumab 20 mg sc. Note: Novartis is not supplying the SARS-CoV-2 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Must have completed a selected Novartis MS study which dosed ofatumumab 20 mg sc every 4 weeks
2. Written informed consent

Exclusion Criteria:

* Emergence of any clinically significant condition/disease during the previous ofatumumab study in which study participation might result in safety risk for the subject
* Subjects with active systemic bacterial, viral or fingal infections, or chronic infection (e.g. AIDS)
* Subjects taking medications prohibited by the protocol
* Pregnant or nursing (lactating) women Other protocol-defined inclusion/exclusion criteria may apply

Vaccination sub-study:

Inclusion criteria

1. Informed consent
2. Actively enrolled in the COMB157G2399 Study
3. 12 weeks of continuous treatment within the COMB157G2399 Study
4. prior vaccination history as per protocol-defined

Exclusion criteria

* known hypersensitivity or history of systemic allergic, neurologic or other reactions to vaccines
* allergies to egg or shellfish
* any safety findings including low IgG/IgM requiring ofatumumab interruption within 12 weeks prior to vaccination sub-study start
* any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 2 weeks of the first vaccination sub-study visit

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1882 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients that experience an adverse event or abnormal laboratory, vital and/or ECG results and positive suicidiality outcomes | Up to 8 years

SECONDARY OUTCOMES:
Number of relapse rates per year | Data from the core studies through the first 5 years in this study.
  Annual Relapse Rate (ARR) time calculated as number of confirmed relapses divided by time in study per year and will also be presented for the entire duration
Patients with confirmed 3 and 6 month disability worsening | During the first 5 years of treatment in the study.
  A confirmed disability worsening is an increase from baseline in Expanded Disability Status Scale (EDSS) score sustained for at last 3, or 6 months EDSS consists of seven functional systems and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, and Cerebral functions (Fatigue contributes).
Patients with confirmed 6, 12, and 24 month disability improvement and improvement during the first 5 years of the study. | During the first 5 years of treatment in the study.
  Confirmed disability improvement is a decrease from baseline in Expanded Disability Status Scale (EDSS) score sustained for at least 6, 12 or 24 months EDSS consists of seven functional systems and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, and Cerebral functions (Fatigue contributes).
Patients with changes in Expanded Disability Status Scale (EDSS) scores | Data from the core studies through the first 5 years in this study, (depending on if first dose was in the core or in this extension study or comparator randomization)
  Score changes in Expanded Disability Status Scale (EDSS) over time EDSS consists of seven functional systems and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, and Cerebral functions (Fatigue contributes).
Changes in and time to 6 month confirmed worsening of Symbol Digit Modalities Test Scores | During the first 5 years of the study.
  Score changes and confirmed 4-point worsening sustained for 6 months in Symbol Digit Modalities Test (SDMT) scores The Symbol Digit Modalities Test is a neuropsychological, timed test for sustained attention and concentration. 3 versions will be used, alternating at each visit where done. The number of correct responses will be counted for the score.
Changes in the Magnetic Resonance Image (MRI) related to brain volume loss | Data from the core studies through the first 5 years in this study.
  Percent change from baseline in brain volume loss (BVL)
Changes in the Magnetic Resonance Image (MRI) related to T2 lesions | Data from the core studies through the first 5 years in this study.
  Number of new or enlarging T2 lesions
Changes in the Magnetic Resonance Image (MRI) related to Gd-enhancing lesions | Data from the core studies through the first 5 years in this study.
  Total number of Gd-enhancing lesions on all MRI scans adjusted for different time of scan versus follow up time in study
Changes in neurofilament light change serum concentration | Data from the core studies through the first 5 years in this study.
  Extent of neurofilament light change concentration in blood NfL is a component of the neuronal cytoskeleton and is released into the cerebrospinal fluid and into subsequently blood following neuro-axonal damage

OTHER OUTCOMES:
Hummoral immune response to TT vaccine | Pre-vaccination, 4 and 8 weeks post-vaccination
  Proportion of subjects with a positive antibody response to TT vaccine measured 4 and 8 weeks after vaccination while treated with ofatumumab
  * 2-fold increase in titer level
  * Tetanus anti-bodies ≥ 0.2 IU/mL
  * Mean titers of anti-tetanus antibody
Hummoral immune response to 13-valent pneumococcal conjugate vaccine (13-PCV) | 4 and 8 weeks
  Proportion of subjects with a positive antibody response against individual anti-pneumococcal antibody serotypes while treated with ofatumumab
  * 2-fold increase in titer level or a > 1 microgram/mL rise in titer compared with pre-immunization titer
  * Positive anti-body response against at least 2 of the 13 pneumococcal antibody serotypes
  * Positive anti-body response against at least 50% of serotypes
  * Mean titers of anti-pneumococcal antibody
Hummoral immune response to 13-PCV boosted eight weeks later by 23-valent pneumococcal polysaccharide vaccine (23-PPV) | Pre-vaccination, 4 and 8 weeks post-vaccination
  Proportion of subjects with a positive antibody response against individual anti-pneumococcal antibody serotypes (23 serotypes to be tested individually) measured 4 and 8 weeks after the booster 23-PPV while the subject continues to be treated with ofatumumab
  * 2-fold increase in titer level or a > 1 microgram/mL rise in titer compared with pre-immunization titer
  * Positive anti-body response against at least 2 of the 23 pneumococcal antibody serotypes
  * Positive anti-body response against at least 50% of serotypes
  * Mean titers of anti-pneumococcal antibody
Humoral immune response to KLH neo-antigen | Pre-administration, 4, 8, 12 weeks after initial administration and 4 weeks after last administration
  Mean titers of anti-KLH antibody measured immediately prior the first administration of KLH and measured immediately prior to the first administration, 4, 8 and 12 weeks after the first administration, and measured 4 weeks post last administration of KLH
Hummoral immune response to 2020-2021 seasonal quadrivalent influenza vaccine | Pre-vaccination and 4 weeks post-vaccination
  Proportion of subjects fulfilling:
  1. Seroconversion: The pre-vaccination HI antibody titer is < 1:10 and the postvaccination measurement is ≥ 1:40 (this applies to subjects with a pre-vaccination HI titer < 1:10), or
  2. Significant increase in HI antibody titer: The pre-vaccination HI antibody titer is ≥ 1:10 and the increase from the pre- to the post-vaccination measurement is ≥ 4-fold (this applies to subjects with a pre-vaccination HI titer ≥ 1:10)
Antibody response rate to TT and influenza vaccination as a function of exposure to ofatumumab | 8 weeks
  Immune response to TT and influenza vaccination

CONTACTS AND LOCATIONS:
Locations (267):
- United States (86):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - North Central Neurology Associates PC, Cullman, Alabama
  - Barrow Neurological Clinics at St Josephs Hospital and MC, Phoenix, Arizona
  - Fullerton Neuro and Headache Ctr, Fullerton, California
  - University of California Davis, Sacramento, California
  - CU Anschutz Med Campus, Aurora, Colorado
  - Mountain Neuro Research Center PC, Basalt, Colorado
  - Alpine Clinical Research Center, Boulder, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Colorado Neurological Research PC, Denver, Colorado
  - University of Colorado Health Neurology, Fort Collins, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Jem Research Institute, Atlantis, Florida
  - Neurology Offices of South Florida PLLC, Delray Beach, Florida
  - Infinity Clinical Research LLC, Hollywood, Florida
  - Homestead Assoc In Research Inc, Homestead, Florida
  - Neurology Associates PA, Maitland, Florida
  - UM Department Of Neurology, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - MS and Neuromuscular Center of Excellence, Oldsmar, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Emerald Coast Neurology, Pensacola, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Negroski Neurology, Sarasota, Florida
  - Roskamp Institute Inc, Sarasota, Florida
  - AMO Corporation, Tallahassee, Florida
  - Clinical Research of West Florida Inc, Tampa, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University Of South Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Velocity Clinical Research, Savannah, Georgia
  - Georgia Neurology and Sleep Medicine Assoc, Suwanee, Georgia
  - Hawaii Pacific Neuroscience LLC, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Consultants in Neurology, Northbrook, Illinois
  - Josephson Wallack Munshower Neurology P.C, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - College Park Family Care Center, Overland Park, Kansas
  - Neuro Medical Clinic of Cenla LLC, Alexandria, Louisiana
  - The Neuromedical Center, Baton Rouge, Louisiana
  - Dragonfly Research LLC, Wellesley Hills, Massachusetts
  - Wayne State University Multiple Sclerosis Clinic, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Vivo Infusion, Plymouth, Minnesota
  - Sharlin Health and Neurology, Ozark, Missouri
  - WA Uni School Of Med, St Louis, Missouri
  - Mercy Research, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Advanced Neurology Specialists, Great Falls, Montana
  - Cleveland Clinic Foundation, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - Ms Ctr Of Northeastern Ny, Latham, New York
  - Asheville Neurology Specialists PA, Asheville, North Carolina
  - The Neurological Institute PA, Charlotte, North Carolina
  - Guilford Neurologic Associate Research, Greensboro, North Carolina
  - Velocity Clinical Research, Raleigh, North Carolina
  - PMG Research of Winston Salem, Winston-Salem, North Carolina
  - Neurology and Neuroscience Assos, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Columbus Neuroscience, Westerville, Ohio
  - Multiple Sclerosis Center of Excellence of OMRF, Oklahoma City, Oklahoma
  - Providence Neurological Services West, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Abington Neurological Associates Ltd, Willow Grove, Pennsylvania
  - Premier Neurology, Greenville, South Carolina
  - BG Neurology, Spartanburg, South Carolina
  - Upstate Clinical Trials LLC, Spartanburg, South Carolina
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Tri State Mountain Neurology, Johnson, Tennessee
  - University of Tennessee Medical Ctr, Knoxville, Tennessee
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Med Research Inc, El Paso, Texas
  - Neurology and Sleep Center, Lubbock, Texas
  - Central TX Neuro Consultants P A, Round Rock, Texas
  - Lonestar Neurology of San Antonio, San Antonio, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Rocky Mountain MS Clinic, Salt Lake City, Utah
  - The University of Utah, Salt Lake City, Utah
  - Sentara Neuroscience Institute, Virginia Beach, Virginia
  - Evergreen Health Multiple Sclerosis Center, Kirkland, Washington
  - MultiCare Research Institute for Research and Innovation, Tacoma, Washington
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - Ascension St Francis Center, Milwaukee, Wisconsin
  - St Luke s Medical Center Aurora, Milwaukee, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, San Miguel de Tucumán
- Australia (3):
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, St Leonards
- Novartis Investigative Site, Vienna, Austria
- Belgium (5):
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Canada (7):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Croatia (3):
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zagreb
- Czechia (8):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Havířov
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Denmark (2):
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Odense C
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (2):
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (7):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (20):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Neuburg A.d. Donau, Bavaria
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Barsinghausen
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (5):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Szeged
- India (8):
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Chandigarh, Punjab
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Howrah, West Bengal
- Israel (4):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Tel Aviv
- Japan (10):
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
- Latvia (2):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Riga
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Chihuahua City
- Netherlands (3):
  - Novartis Investigative Site, Sittard-Geleen, Limburg
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Rotterdam, South Holland
- Novartis Investigative Site, Drammen, Norway
- Peru (3):
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Lima
- Poland (11):
  - Novartis Investigative Site, Bydgoszcz, Woj Kujawsko Pomorskie
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Glogow Wielkopolski
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
- Portugal (7):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Loures
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Santa Maria da Feira
- Russia (11):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saransk
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (5):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Trnava
- South Africa (2):
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Rosebank
- Spain (15):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Donostia / San Sebastian, Gipuzkoa
  - Novartis Investigative Site, Salt, Girona
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Castilleja de la Cuesta, Sevilla
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lugano
- Novartis Investigative Site, Tainan, Taiwan
- Novartis Investigative Site, Khon Kaen, THA, Thailand
- Turkey (Türkiye) (11):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Istanbul, Bakirkoy
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Izmir, Karsiyaka
  - Novartis Investigative Site, Trabzon, Ortahisar
  - Novartis Investigative Site, Istanbul, Sancaktepe
  - Novartis Investigative Site, Istanbul, Sultangazi
  - Novartis Investigative Site, Mersin, Yenisehir
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
- United Kingdom (5):
  - Novartis Investigative Site, Luton, Beds
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hauser SL, Cohen JA, de Seze J, Meuth SG, Giacomini PS, Nakahara J, Oreja-Guevara C, Robertson D, Wray S, Bhatt A, Hu X, Xi J, Piccolo R, Jehl V, Sullivan R, Boer I, Wiendl H, Kappos L. Five-Year Safety and Efficacy Outcomes with Ofatumumab in Patients with Relapsing Multiple Sclerosis. Neurol Ther. 2025 Oct;14(5):1975-1992. doi: 10.1007/s40120-025-00784-0. Epub 2025 Jul 13. PMID 40652442
- [Derived] Hauser SL, Zielman R, Das Gupta A, Xi J, Stoneman D, Karlsson G, Robertson D, Cohen JA, Kappos L. Efficacy and safety of four-year ofatumumab treatment in relapsing multiple sclerosis: The ALITHIOS open-label extension. Mult Scler. 2023 Oct;29(11-12):1452-1464. doi: 10.1177/13524585231195346. Epub 2023 Sep 11. PMID 37691530